CLINICAL TRIAL: NCT06709105
Title: The Effect of Kinesiotaping on Clinical Parameters in Pregnant Women With Mechanical Low Back Pain
Brief Title: The Effect of Kinesiotaping in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Muhammet Sahin Elbasti, Head of Physical Medicine and Rehabilitation Departmant, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 192
Record Dates: First submitted 2024-11-21; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: KINESIOTAPING
Keywords: Kinesiotaping; Low Back Pain; Pregnancy
MeSH Terms: conditions — Low Back Pain | interventions — Athletic Tape; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotape application (Experimental): The application was performed using 5 cm x 5 m kinesio tape material. After preparing the standing patient in terms of clothing and skin readiness, the patient was asked to lean forward. To adhere the tape to the right paravertebral region, the lower end of the tape was first adhered 7 cm below the sacroiliac joint at the level of the paravertebral muscles. Then, while the patient was leaning forward, a slight rotation to the left was requested, and in this position, the tape was adhered upwards along the paravertebral muscles without any tension. When applying the tape to the left paravertebral region, the same procedure was mirrored as on the right, with the tape again applied without any tension. The third tape was applied while the patient was standing upright and leaning slightly forward, placed over the sacroiliac joints and parallel to the floor, stretching the tape by 25%.
  Interventions: Other: Kinesiotape
- Sham group (Sham Comparator): Sham Kinesio taping was applied to the patients in the control group. In this sham protocol, Kinesio bands were attached between the 12th rib on both sides and the corresponding sacroiliac joint, passing over the paravertebral muscles without employing any specific banding technique. The third tape was adhered between both sacroiliac joints, also without any adhesive technique. Patients were inquired about any discomfort and informed that the tapes would remain in place until the second session.
  Interventions: Other: Sham (no implant)

INTERVENTIONS:
Other: Kinesiotape — The application was performed using 5 cm x 5 m kinesio tape material. After preparing the standing patient in terms of clothing and skin readiness, the patient was asked to lean forward. To adhere the tape to the right paravertebral region, the lower end of the tape was first adhered 7 cm below the sacroiliac joint at the level of the paravertebral muscles. Then, while the patient was leaning forward, a slight rotation to the left was requested, and in this position, the tape was adhered upwards along the paravertebral muscles without any tension. When applying the tape to the left paravertebral region, the same procedure was mirrored as on the right, with the tape again applied without any tension. The third tape was applied while the patient was standing upright and leaning slightly forward, placed over the sacroiliac joints and parallel to the floor, stretching the tape by 25%.
  Arms: Kinesiotape application
Other: Sham (no implant) — Sham Kinesio taping was applied to the patients in the control group. In this sham protocol, Kinesio bands were attached between the 12th rib on both sides and the corresponding sacroiliac joint, passing over the paravertebral muscles without employing any specific banding technique. The third tape was adhered between both sacroiliac joints, also without any adhesive technique. Patients were inquired about any discomfort and informed that the tapes would remain in place until the second session.
  Arms: Sham group

SUMMARY:
The aim of this study is to examine the effect of an exercise program combined with Kinesio Taping (KT) and sham KT on clinical parameters in pregnant women with low back pain. A total of 40 participants were included in the study, 20 in the experimental and 20 in the control groups. Visual Analog Scale (VAS), Roland Morris Quality of Life Questionnaire and Pittsburgh Sleep Quality Index were used as data collection tools. The experimental group received KT and an exercise program, while the control group received sham KT and exercise program.

DETAILED DESCRIPTION:
Lumbar-sacral spinal pain is a medical and socioeconomic problem affecting approximately 80% of the population. Pregnancy predisposes women to this pain. The most well-known cause of low back pain during pregnancy is an increase in lumbar lordosis, a lordotic syndrome that develops rapidly due to the pregnant uterus and maternal weight gain. This lordotic posture and the related change in load distribution, along with lengthening abdominal muscles and shortening lumbar muscles, create a mechanical disadvantage. The aim of this study is to examine the effect of an exercise program combined with Kinesio Taping (KT) and sham KT on clinical parameters in pregnant women with low back pain. A total of 40 participants were included in the study, 20 in the experimental and 20 in the control groups. Visual Analog Scale (VAS), Roland Morris Quality of Life Questionnaire and Pittsburgh Sleep Quality Index were used as data collection tools. The experimental group received KT and an exercise program, while the control group received sham KT and exercise program.

ELIGIBILITY:
Inclusion Criteria:

* 20-32-week pregnant women without neurologic deficits
* Females with mechanical low back pain
* VAS of at least 3

Exclusion Criteria:

* High-risk pregnant women with twin pregnancy
* Placenta previa
* Pre-eclampsia
* Threatened preterm delivery
* Orthopedic and rheumatologic diseases
* Radiculopathy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | up to 30 minutes
  The Visual Analogue Scale (VAS) has been widely used in numerous studies to assess the intensity of pain and is considered a reliable and valid tool. It measures subjectively perceived pain on a scale resembling a 0-10 cm ruler, with one end representing no pain and the other indicating the most severe pain.

SECONDARY OUTCOMES:
Pittsburgh sleep quality index | up to 30 minutes
  The sleep quality scale, developed by Buysse et al., had its Turkish reliability and validity study conducted by Agargün et al. (1996) This scale assesses an individual's sleep quality over the past month and includes 24 items. Of these, 19 are self-reported questions answered by the individual, and five are answered by a roommate or spouse.

CONTACTS AND LOCATIONS:
Locations (1):
- Muhammet Şahin Elbastı, Elâzığ, Firat University, Turkey (Türkiye)